CLINICAL TRIAL: NCT06712381
Title: Carac & PDT Combination in the Treatment Of Actinic Keratoses
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Skin Laser & Surgery Specialists (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLSS-DG08
Record Dates: First submitted 2016-04-19; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Actinic Keratoses
Keywords: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic | interventions — Fluorouracil; Photochemotherapy; 1-phenyl-3,3-dimethyltriazene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1 (Active Comparator): Carac
  Interventions: Drug: Fluorouracil
- 2 (Active Comparator): Photodynamic Therapy
  Interventions: Procedure: Photodynamic therapy
- 3 (Active Comparator): Carac combined with Photodynamic Therapy
  Interventions: Procedure: Carac in combination with PDT

INTERVENTIONS:
Drug: Fluorouracil — Carac (fluorouracil) Cream, 0.5% is used by adults to treat skin conditions on the face and front part of the scalp called solar keratosis or actinic keratosis.
  Other Names: Carac
  Arms: 1
Procedure: Photodynamic therapy — Photodynamic therapy (PDT) is a procedure that uses a photosensitizing drug to apply light therapy selectively to target pre-skin cancer, acne and sun damage.
  Arms: 2
Procedure: Carac in combination with PDT
  Arms: 3

SUMMARY:
To demonstrate if Carac treatment after PDT treatment of actinic keratoses leads to superior clinical improvement when compared to Carac or PDT treatment alone. This will be done by manual counts and through photography.

DETAILED DESCRIPTION:
Carac has been shown to be highly effective for the treatment of actinic keratoses. Photodynamic Therapy (PDT) has also been shown to be highly effective for the treatment of actinic keratoses. Both treatments are FDA approved. The mechanism of action of each therapy is different. In general a more vigorous, but less cosmetically acceptable appearance is seen after Carac treatment as compared to PDT treatment. The purposes of this study are to determine 1) If the use of Carac, followed by PDT treatment, of actinic keratoses leads to an enhanced clinical improvement as compared to PDT treatment alone; 2) If the cosmetic appearance of the skin during Carac is improved with PDT pre-treatment; 3) Evaluate histologic changes induced by combined Carac/PDT treatment as compared to Carac treatment alone and PDT treatment alone.;4) Evaluate safety of treatments in terms of potential for infection and scarring

ELIGIBILITY:
Inclusion Criteria:

* Males/females,, aged 40-70
* Must have 5 or more documented facial/anterior scalp actinic keratoses
* Read, understood, and signed informed consent form
* Willing and able to comply with all follow-up requirements

Exclusion Criteria:

* Previous treatment of facial keratoses with any modality of treatment within 3 months of study enrollment
* Contraindications to the use of either Carac and/or PDT treatment
* Exclusion of biopsy proven skin cancer in the area
* Active infections or dermatitis in the treatment area

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Reduction of Actinic Keratoses | Outcomes are assessed at 3 months
  The objective of this study is to demonstrate if Carac treatment after PDT treatment of actinic keratoses leads to superior clinical improvement when compared to Carac or PDT treatment alone based on a manual lesion count.

SECONDARY OUTCOMES:
Photographic Improvement of Actinic Keratoses | Outcomes are assessed at 3 months
  The objective of this study is to demonstrate if Carac treatment after PDT treatment of actinic keratoses leads to superior clinical improvement when compared to Carac or PDT treatment alone based on a photographic improvement using the Actinic Keratosis-Field Assessment Scale.